CLINICAL TRIAL: NCT04228913
Title: Comparison of Postoperative Pain Intensity After Three Different Obturation Techniques: A Randomized Clinical Trial
Brief Title: Effect of Different Obturation Techniques on Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Hicran Dönmez Özkan, Assistant Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ADÜDHF 2017/021
Record Dates: First submitted 2020-01-07; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Pain, Postoperative; Pain; Endodontic Inflammation
Keywords: cold lateral condensation; Postoperative Pain; GuttaCore; GuttaFlow 2; Obturation Techniques
MeSH Terms: conditions — Pain, Postoperative; Pain; Pulpitis

STUDY DESIGN:
Intervention Model Description: Single (Participant)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ah plus (Other): The root canals obturated with Ah plus root canal sealer (Dentsply, Sirona) and gutta-percha cones with cold lateral condensation technique.
  Interventions: Other: Root Canal Obturation Technique
- ROEKO GuttaFlow® 2 (Other): The root canals obturated with GuttaFlow 2 root canal sealer (Coltene,Whaledent) and single tapered gutta-percha cone with cold free flow compaction technique.
  Interventions: Other: Root Canal Obturation Technique
- GuttaCore Obturators (Other): The root canals obturated with GuttaCore obturators (Dentsply,Sirona) and Ah plus root canal sealer with thermoplasticized solid-core carrier technique
  Interventions: Other: Root Canal Obturation Technique

INTERVENTIONS:
Other: Root Canal Obturation Technique — This study aims to compare the effects of three different obturation techniques(cold lateral condensation,thermoplasticized solid-core carrier method, cold free flow compaction technique) on postoperative pain following the endodontic therapy

SUMMARY:
This study evaluated the postoperative pain after the endodontic treatment by using three different obturation techniques. ( Cold lateral condensation (CLC), thermoplasticized solid-core carrier method (GuttaCore) and cold free-flow compation tecnique ( GuttaFlow2))

ELIGIBILITY:
Inclusion Criteria:

1. Participants between 18 - 72 years of ages,

2 Good oral hygiene,

3. Have not taken any analgesic in the last 7 days,

4. Have not taken any antibiotics in the last 7 days,

5. Positive response to both cold test (EndoIce; Coltene/Whaledent Inc, Cuyahoga ),

6. Patients diagnosed with asymptomatic irreversible pulpitis with his/her single-rooted teeth caused by a deep carious lesion,

7. Patients have single-rooted teeth requiring endodontic treatment according to the pre-prosthetic reason,

8.The presence of profusely pulp bleeding with a thick consistency, which is exposed during caries removing.

9. The periapical region was healthy in radiographic diagnosis.

Exclusion Criteria:

1. Patients who refuse to participate in this study,
2. Medically compromised patients (with immunosuppressive/systemic diseases, patients on medications),
3. Devital teeth that have no response to pulp test,
4. The presence of advanced periodontal disease (probing depth > 4 mm),
5. The presence of open apex,
6. The presence of calcification,
7. The presence of resorption,
8. Patients who had multiple teeth requiring endodontic treatment,
9. Patients with allergic sensitivity to materials and agents that should be used during the root canal treatment,
10. Allergic sensitivity to local anesthetics,
11. Patients who had systemic or allergic sensitivity for the NSAIDs,
12. Pregnant participants or participants in the lactation period,
13. Teeth cannot be applied to a rubber-dam.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Pain level comparison after root canal obturation with three different obturation technique:: VAS (Visual Analogue Scale) at 6th hours. | 6th hours.
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different obturation technique.: VAS (Visual Analogue Scale) at 12th hours. | 12th hours.
  ased on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different obturation technique.: VAS (Visual Analogue Scale) at 24th hours | 24th hours.
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different obturation technique.: VAS (Visual Analogue Scale) at 2nd days. | 2nd days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different obturation technique.: VAS (Visual Analogue Scale) at 3th days. | 3th days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different obturation technique.: VAS (Visual Analogue Scale) at 4th days. | 4th days.
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different obturation technique.: VAS (Visual Analogue Scale) at 5th days. | 5th days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different obturation technique.: VAS (Visual Analogue Scale) at 6th days. | 6th days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after root canal obturation with three different obturation technique.: VAS (Visual Analogue Scale) at 7th days. | 7th days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.

SECONDARY OUTCOMES:
Analgesic intake comparison after root canal obturation with three different obturation technique at 6th hours | 6th hours.
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different obturation technique at 12th hours | 12th hours
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different obturation technique at 24th hours | 24th hours.
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different obturation technique at 2nd days | 2nd days
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different obturation technique at 3th days | 3th days
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different obturation technique at 4th days | 4 th days
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different obturation technique at 5th days | 5th days
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different obturation technique at 6th days | 6th days
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"
Analgesic intake comparison after root canal obturation with three different obturation technique at 7th days | 7th days.
  The patients were asked to choose one of the three options: "0: No pain, or no pain which does not require the use of analgesics", "1: Moderate pain which can be controlled very well by the use of analgesics and does not affect daily activities or sleep", "2: Daily activities Unbearable pain that cannot be controlled by the use of analgesics"

CONTACTS AND LOCATIONS:
Overall Officials: Hicran Dönmez Özkan, Study Director — Adnan Menderes University, Faculty of Dentistry
Locations (1):
- Hicran Dönmez Özkan, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alonso-Ezpeleta LO, Gasco-Garcia C, Castellanos-Cosano L, Martin-Gonzalez J, Lopez-Frias FJ, Segura-Egea JJ. Postoperative pain after one-visit root-canal treatment on teeth with vital pulps: comparison of three different obturation techniques. Med Oral Patol Oral Cir Bucal. 2012 Jul 1;17(4):e721-7. doi: 10.4317/medoral.17898. PMID 22322522
- [Background] Su Y, Wang C, Ye L. Healing rate and post-obturation pain of single- versus multiple-visit endodontic treatment for infected root canals: a systematic review. J Endod. 2011 Feb;37(2):125-32. doi: 10.1016/j.joen.2010.09.005. Epub 2010 Nov 12. PMID 21238790
- [Result] Graunaite I, Skucaite N, Lodiene G, Agentiene I, Machiulskiene V. Effect of Resin-based and Bioceramic Root Canal Sealers on Postoperative Pain: A Split-mouth Randomized Controlled Trial. J Endod. 2018 May;44(5):689-693. doi: 10.1016/j.joen.2018.02.010. Epub 2018 Mar 20. PMID 29571915
- [Derived] Kocer A, Donmez Ozkan H, Turk T. Postoperative pain intensity and incidence following single visit root canal treatment with different obturation techniques: a randomized clinical trial. PeerJ. 2022 Jul 27;10:e13756. doi: 10.7717/peerj.13756. eCollection 2022. PMID 35915749